CLINICAL TRIAL: NCT00244127
Title: Cyclophosphamide, Oncovin, Myocet, Prednisone and Rituximab (R-COMP) in the Treatment of Elderly Patients With Aggressive NHL.
Brief Title: Open Label, Single Arm, Phase II Study Using R-COMP in Elderly Patients With Aggressive NHL.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zeneus Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Myocet 018; The MYOCAN Study
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2005-10

CONDITIONS: Aggressive Non-Hodgkin's Lymphoma in the Elderly.
MeSH Terms: interventions — Cyclophosphamide; Vincristine; Doxorubicin; Prednisone; Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide, oncovin, myocet, prednisone & rituximab (R-COMP)

SUMMARY:
To evaluate the safety and efficacy of R-COMP in elderly patients with advanced aggressive NHL. Myocet (non-pegylated liposomal doxorubicin) replaces conventional doxorubicin in the R-CHOP regimen.

DETAILED DESCRIPTION:
To evaluate the duration of remission, disease free survival and 2-year survival of R-COMP in first line therapy of elderly patients with advanced aggressive NHL.

To evaluate the tolerability of R-COMP in first line therapy of elderly patients with advanced aggressive NHL.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse Large B-Cell Lymphoma (DLBCL), and their morphologic variants and subtypes, i.e. Centroblastic lymphoma, Immunoblastic lymphoma, T-cell rich/B-cell lymphoma, anaplastic large B-cell lymphoma, mediastinal (thymic) large B-cell lymphoma;
* Primary diffuse large B-cell lymphoma of MALT (incorrectly defined as high-grade MALT lymphoma);
* Marginal zone B-cell lymphoma with coexisting areas of DLBCL;
* Age of ≥60 years;
* Clinical stage at diagnosis: I A bulky - IV B;
* CD20 positivity;
* Serum negativity for HbsAg and HCV except for those with no sign of active viral replication, assessed by HCV-RNA copies;
* Absolute neutrophil count (ANC) ≥1.5x109/L, and platelet count ≥100x109/L (unless both are attributed directly to bone marrow involvement by lymphoma or auto-immune disease secondary to lymphoma);
* Serum creatinine ≤130μM/L, serum bilirubin ≤2.5xULN aspartate amino-transferase (AST/GOT), ≤2.5xULN alanine amino-transferase (ALT/GPT) ≤2.5xULN, and alkaline phosphatase ≤4 times the upper limit of normal (unless the increase is attributed directly to the presence of tumour by the Investigator)
* Left ventricular ejection fraction (LVEF) ≥50%;
* ECOG performance status 0-2;
* At least one measurable lesion is mandatory;
* Written informed consent given at time of registration;
* Males and females (both males and females of childbearing potential must agree to use adequate contraception for the duration, and for 3 months after the completion, of the treatment).

Exclusion Criteria:

* Clinical stage I non-bulky, or CS IIA with less than three sites of disease involved (patients with stage IIB are eligible, regardless of the number of sites involved);
* Tumour involvement of CNS;
* Indolent lymphoma transformed in more aggressive histological type, even if never previously treated;
* Mantle Cell Lymphoma, Peripheral T cell Lymphoma and their variants;
* Aggressive non-Hodgkin's lymphoma in transplanted patient;
* Clinically significant secondary cardiovascular disease, e.g. uncontrolled hypertension, (resting diastolic blood pressure >115 mmHg), uncontrolled multifocal cardiac arrhythmias, symptomatic angina pectoris or congestive cardiac failure NYHA class III-IV;
* Evidence of any severe active acute or chronic infection;
* Concurrent malignancy or history of other malignancy, except basal cell carcinoma of the skin (BCC) and in-situ cervical carcinoma (CIN) / Myelodysplastic syndrome;
* HbsAg, HIV-positive, or HCV-RNA-positive patients;
* Inability to comply with study procedures;
* Prior CNS lymphoma;
* Prior radiation to non-CNS lymphoma mass(es) as a treatment for lymphomas;
* History of allergic reaction to anthracyclines, eggs, and egg products or known sensitivities, or history of unusual reaction, to other components of, or treatments similar to, the investigational treatment regimen;
* Presence of other medication that may interfere with study treatment or the action of the investigational product or confuse the assessment of study results
* Pregnant women or nursing mothers;
* Participation in an investigational drug study within 4 weeks prior to study entry.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75
Dates: Start 2002-10

PRIMARY OUTCOMES:
Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, Principal Investigator — Universita Degli Studi di Modena
Locations (5):
- Paris, France
- Berlin, Germany
- Universita Degli Studi Di Modena AZ Ospedaliere Policlinico, Modena, Italy
- Barcelona, Spain
- Leicester, United Kingdom